CLINICAL TRIAL: NCT01033864
Title: Comparison of Pharmocokinetics of Mycophenolate Mofetil and Enteric Coated Mycophenolate Sodium in Calcineurininhibitor-free Treated Patients After Renal Transplantation
Brief Title: A Pharmacokinetic Study of CellCept (Mycophenolate Mofetil) Versus Mycophenolate Sodium in Kidney Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22641; 2009-012355-15
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Prednisone

ARMS (2):
- MMF, Prednisone (Experimental): Participants received mycophenolate mofetil (MMF) orally (PO) at a dose of 1 gram per day (g/day) twice daily (BID), and prednisone, PO, up to 5 milligrams per day (mg/day) for at least 1 month.
  Interventions: Drug: MMF; Drug: Prednisone
- EC-MPS (Active Comparator): Participants received mycophenolate sodium (EC-MPS), PO, at a dose of 720 mg/day BID, and prednisone PO up to 5 mg/day for at least 1 month.
  Interventions: Drug: EC-MPS; Drug: Prednisone

INTERVENTIONS:
Drug: MMF — 1 g per day b.i.d. p.o. for at least 1 month
  Other Names: CellCept; mycophenolate mofetil
  Arms: MMF, Prednisone
Drug: EC-MPS — 720 mg b.i.d. p.o. for at least 1 month
  Other Names: mycophenolate sodium
  Arms: EC-MPS
Drug: Prednisone — 5 mg per day p.o.

SUMMARY:
This open-label, 2-arm study will compare the pharmacokinetics of CellCept and mycophenolate sodium in kidney transplanted patients on a calcineurininhibitor-free mycophenolic acid-based therapy. On the study day patients will take their prescribed medication (either CellCept or mycophenolate sodium). Blood samples will be drawn directly before and at intervals up to 12 hours after intake of the study medication. Anticipated time on study treatment is 12 hours and target sample size is 24.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* kidney transplantation >/=6 months ago
* on mycophenolic acid-based, calcineurininhibitor-free therapy for >/=3 months, >/=1 month on stable dose
* co-therapy with 5mg prednisone for >/=1 month

Exclusion Criteria:

* active gastrointestinal ulcus
* severe diarrhea od gastrointestinal disease
* severe impairment of renal function
* current malignancy
* Lesch-Nyhan- or Kelley-Seegmiller-Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Frankfurt am Main, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Mofetil (MMF)/Prednisone: Participants were administered MMF tablets or capsules, orally (PO), at a dose prescribed by their physician and prednisone up to 5 milligrams (mg) PO on Day 1.
- Enteric-coated Mycophenolate Sodium (EC-MPS)/Prednisone: Participants were administered EC-MPS tablets, PO, at a dose prescribed by their physician and prednisone up to 5 mg PO on Day 1.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil (MMF)/Prednisone | Enteric-coated Mycophenolate Sodium (EC-MPS)/Prednisone
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The pharmacokinetic (PK) population included all randomized participants.
Groups:
- MMF/Prednisone: Participants were administered MMF tablets or capsules, PO, at a dose prescribed by their physician and prednisone up to 5 mg PO on Day 1.
- EC-MPS/Prednisone: Participants were administered EC-MPS tablets, PO, at a dose prescribed by their physician and prednisone up to 5 mg PO on Day 1.
- Total: Total of all reporting groups
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.06) [42 to 76] | 58.0 (8.04) [49 to 74] | 59.8 (9.68) [NA to NA]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Pre-dose Trough Concentration (C0)
Description: The mean mycophenolic acid (MPA) concentration in plasma was determined (in milligrams per liter [mg/L]) from blood samples collected predose (immediately before receiving study treatment).
Time Frame: Day 1 predose
Population: Pharmacokinetic (PK) population: all participants who took study drug and for whom all defined blood samples at the planned sampling time points were available.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone
Number analyzed (Participants) | 12 | 11
mg/L | 2.387 (1.1327) | 2.944 (2.2103)
Statistical Analysis 1: Comparison: MMF/Prednisone vs EC-MPS/Prednisone; Test type: Superiority or Other; p = 0.8055, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Dose-Normalized C0
Description: Dose normalized C0 was determined (in mg/L) from blood samples collected predose. Both MMF and EC-MPS doses were normalized to a standard dose of 1 g MMF or 720 mg EC-MPS, respectively. The dose normalization was calculated as follows:
  For the MMF group: Dose normalized C0 equals (=) C0 divided by (/) (actual dose taken/1000) For the EC-MPS group: Dose normalized C0 = C0 / (actual dose taken/720)
Time Frame: Day 1 predose
Population: PK population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone
Number analyzed (Participants) | 12 | 11
mg/L | 2.962 (1.4439) | 4.658 (3.1121)
Statistical Analysis 1: Comparison: MMF/Prednisone vs EC-MPS/Prednisone; Test type: Superiority or Other; p = 0.2548, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Minimum Plasma Concentration (Cmin)
Description: The mean minimum MPA concentration in plasma was determined (in mg/L) from blood samples collected predose and postdose on Day 1.
Time Frame: Day 1 predose and postdose at 30 and 60 minutes and 2, 3, 4, 5, 6, 8 10 and 12 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone
Number analyzed (Participants) | 12 | 11
mg/L | 1.385 (0.6061) | 1.620 (0.6632)
Statistical Analysis 1: Comparison: MMF/Prednisone vs EC-MPS/Prednisone; Test type: Superiority or Other; p = 0.4417, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Dose-Normalized Cmin
Description: Dose-normalized Cmin was determined (in mg/L) from blood samples collected predose and postdose. Both MMF and EC-MPS doses were normalized to a standard dose of 1 g MMF or 720 mg EC-MPS, respectively. The dose normalization was calculated as follows:
  For the MMF group: Dose normalized Cmin = Cmin/ (actual dose taken/1000) For the EC-MPS group: Dose normalized Cmin = Cmin / (actual dose taken/720)
Time Frame: Day 1 predose and postdose at 30 and 60 minutes and 2, 3, 4, 5, 6, 8 10 and 12 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone
Number analyzed (Participants) | 12 | 11
mg/L | 1.702 (0.8018) | 2.613 (1.0291)
Statistical Analysis 1: Comparison: MMF/Prednisone vs EC-MPS/Prednisone; Test type: Superiority or Other; p = 0.0455, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The mean maximum MPA concentration in plasma was determined (in mg/L) in blood samples collected predose and postdose on Day 1.
Time Frame: Day 1 predose and postdose at 30 and 60 minutes and 2, 3, 4, 5, 6, 8 10 and 12 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone
Number analyzed (Participants) | 12 | 11
mg/L | 15.385 (5.2320) | 17.827 (4.2898)
Statistical Analysis 1: Comparison: MMF/Prednisone vs EC-MPS/Prednisone; Test type: Superiority or Other; p = 0.2300, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Dose-Normalized Cmax (mg/L)
Description: Dose-normalized Cmax in plasma was determined (in mg/L) from blood samples collected predose and postdose on Day 1. Both MMF and EC-MPS doses were normalized to a standard dose of 1 g MMF or 720 mg EC-MPS, respectively. The dose normalization was calculated as follows:
  For the MMF group: Dose normalized Cmax = Cmax / (actual dose taken/1000) For the EC-MPS group: Dose normalized Cmax = Cmax / (actual dose taken/720)
Time Frame: Day 1 predose and postdose at 30 and 60 minutes and 2, 3, 4, 5, 6, 8 10 and 12 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone
Number analyzed (Participants) | 12 | 11
mg/L | 18.402 (5.4349) | 29.996 (11.3229)
Statistical Analysis 1: Comparison: MMF/Prednisone vs EC-MPS/Prednisone; Test type: Superiority or Other; p = 0.0106, Wilcoxon (Mann-Whitney)

7. Primary Outcome: MPA Area Under the Curve From 0 to 12 Hours (AUC0-12)
Description: The mean MPA AUC0-12 in plasma was determined (in mg multiplied by hours, per Liter [mg*h/L]) from blood samples collected predose and postdose on Day 1.
Time Frame: Day 1 predose and postdose at 30 and 60 minutes and 2, 3, 4, 5, 6, 8 10 and 12 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone
Number analyzed (Participants) | 12 | 11
mg*h/L | 50.36348 (15.423230) | 57.06682 (10.965285)
Statistical Analysis 1: Comparison: MMF/Prednisone vs EC-MPS/Prednisone; Test type: Superiority or Other; p = 0.3401, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Dose-Normalized MPA AUC0-12
Description: Dose-normalized MPA AUC0-12 in plasma was determined (mg*h/L) from blood samples collected predose and postdose on Day 1. Both MMF and EC-MPS doses were normalized to a standard dose of 1 g MMF or 720 mg EC-MPS, respectively. The dose normalization was calculated as follows:
  For the MMF group: Dose normalized MPA AUC = MPA AUC / (actual dose taken/1000) For the EC-MPS group: Dose normalized MPA AUC = MPA AUC / (actual dose taken/720)
Time Frame: Day 1 predose and postdose at 30 and 60 minutes and 2, 3, 4, 5, 6, 8 10 and 12 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone
Number analyzed (Participants) | 12 | 11
mg*h/L | 61.53862 (21.003959) | 94.65765 (29.307839)
Statistical Analysis 1: Comparison: MMF/Prednisone vs EC-MPS/Prednisone; Test type: Superiority or Other; p = 0.0074, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Percentage of Participants By Time to Maximum Plasma Concentration (Tmax)
Time Frame: Day 1 predose and postdose at 30 and 60 minutes and 2, 3, 4, 5, 6, 8 10 and 12 hours
Population: PK population
Measure: Number; unit: percentage of participants
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone
Number analyzed (Participants) | 12 | 11
percentage of participants
  Tmax equals (=) 0.5333 hours (hrs) | 16.7 | 0.0
  Tmax=0.6000 hrs | 16.7 | 0.0
  Tmax=0.7333 hrs | 16.7 | 0.0
  Tmax=0.7667 hrs | 8.3 | 0.0
  Tmax=1.0667 hrs | 8.3 | 9.1
  Tmax=1.0833 hrs | 16.7 | 0.0
  Tmax=1.1167 hrs | 8.3 | 0.0
  Tmax=1.2167 hrs | 8.3 | 0.0
  Tmax=2.0167 hrs | 0.0 | 9.1
  Tmax=2.0833 hrs | 0.0 | 18.2
  Tmax=2.1000 hrs | 0.0 | 9.1
  Tmax=2.1167 hrs | 0.0 | 27.3
  Tmax=2.1667 hrs | 0.0 | 9.1
  Tmax=3.1167 hrs | 0.0 | 9.1
  Tmax=3.1833 hrs | 0.0 | 9.1
Statistical Analysis 1: Comparison: MMF/Prednisone vs EC-MPS/Prednisone; Test type: Superiority or Other; p = 0.0002, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Regression Coefficients For Participants Receiving MMF
Description: The estimated regression coefficients for participants who received MMF presented in milligrams per liter (mg/L).
Time Frame: Day 1 at 30 minutes and 1 and 2 hours postdose
Population: PK population. Only participants in the MMF/Prednisone group were assessed for this outcome measure, n=12.
Measure: Number; unit: mg/L
Arm/Group | MMF/Prednisone
Number analyzed (Participants) | 12
mg/L
  Intercept | 2.17192
  Concentration at 30 minutes (C0.5) | 0.74031
  Concentration at 1 hour (C1) | 1.89323
  Concentration at 2 hours (C2) | 2.85923

ADVERSE EVENTS:
Time Frame: The observational period, approximately 13 hours.
Description: All randomized participants were included in the safety analysis.
Arm/Group | MMF/Prednisone | EC-MPS/Prednisone
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.